CLINICAL TRIAL: NCT05456347
Title: A Randomized Study to Investigate the Effect of a Low-calorie and High-protein Diet Specially Rich in Animal Protein Compared to a Low-calorie and High-protein Diet Specially Rich in Plant Protein on Glucose Metabolism in Subjects With Prediabetes or Type 2 Diabetes and Overweight or Obesity.
Brief Title: Effect of a Low-calorie and High-protein Diet Specially Rich in Animal Protein Compared to a Low-calorie and High-protein Diet Specially Rich in Plant Protein on Glucose Metabolism in Subjects With Prediabetes or Type 2 Diabetes and Overweight or Obesity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Rocio Mateo-Gallego, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI19/485
Record Dates: First submitted 2022-07-01; First posted 2022-07-13 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus, Type 2; Overweight and Obesity; PreDiabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Prediabetic State | interventions — Diet, High-Protein

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-protein animal diet. (Experimental): Low-calorie and high-protein diet (35% of total calories), mostly of protein coming from animal sources (75% of total protein).
  Interventions: Behavioral: Low-calorie and high-protein diet with the majority of protein coming from animal sources.
- High-protein vegetal diet. (Experimental): Low-calorie and high-protein diet (35% of total calories), mostly of protein coming from plant sources (75% of total protein).
  Interventions: Behavioral: Low-calorie and high-protein diet with the majority of protein coming from plant sources.

INTERVENTIONS:
Behavioral: Low-calorie and high-protein diet with the majority of protein coming from animal sources. — Diet was prescribed to the participant and menus and recipes were also provided.
  Arms: High-protein animal diet.
Behavioral: Low-calorie and high-protein diet with the majority of protein coming from plant sources. — Diet was prescribed to the participant and menus and recipes were also provided.
  Arms: High-protein vegetal diet.

SUMMARY:
The aim of the study is to explore the effect of a low-calorie diet rich in protein (with a content of 35% of the total calories of the diet), mostly coming from animal sources (75% of total protein), compared to a hypocaloric diet rich in protein (with a content of 35% of the total calories of the diet), mostly coming from plant sources (75% of total proteins), in subjects with prediabetes or type 2 diabetes and overweight or obesity, on body composition, glucose and lipid metabolisms, after 6 months of intervention.

To achieve the objective, a nutritional intervention study is carried out by randomizing participants to: a) a hypocaloric and high-protein diet (35% of total calories), mostly of them coming from animal sources (75% of total protein); b) a hypocaloric and high-protein diet (35% of total calories), mostly of them coming from plant sources (75% of total protein). The study has a total duration of 6 months and include the assessment of clinical, anthropometric, biochemical and lifestyle parameters, at the beginning of the study and after 3 and 6 months of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80.
* BMI between 27.5 kg/m2 and 40 kg/m2.
* Diagnosed as prediabetes or type 2 diabetes according to ADA criteria.
* Informed consent to be signed.

Exclusion Criteria:

* Taking antidiabetic drugs (except for metformin with stable dose in the previous 6 months).
* Taking lipid-lowering drugs in unstable dose in the previous 2 months.
* Taking functional foods (i.e. sterols enriched food) or any other dietary supplement with a significant effect on lipid and glucose metabolism and body weight.
* Uncontrolled type 2 diabetes (i.e. glycated hemoglobin over 8%)
* Any disease that could affect study results (i.e. uncontrolled hypothyroidism).
* Alcohol intake over 30 g/day.
* Pregnancy or breastfeeding.
* Any other condition that investigators consider that could interfere with study outcomes.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Glucose change. | After 3 and 6 months of intervention.
  Glucose change assessed by difference in fasting glucose concentration (mg/dL and %) comparing 3 and 6 months visits with respect to baseline.
Glycated hemoglobin change. | After 3 and 6 months of intervention.
  Glycated hemoglobin change assessed by difference in glycated hemoglobin concentration (%) comparing 3 and 6 months visits with respect to baseline.
Insulin change. | After 3 and 6 months of intervention.
  Insulin change assessed by difference in fasting insulin concentration (UI/mL and %) comparing 3 and 6 months visits with respect to baseline.
HOMA-IR change. | After 3 and 6 months of intervention.
  HOMA-IR change assessed by difference in HOMA-IR concentration (absolute units and %) comparing 3 and 6 months visits with respect to baseline. HOMA-IR is calculated by calculating: [(fasting glucose (mg/dL) x 0,0555) x fasting insulin (UI/ml)] ÷ 22,5.
Body fat mass change. | After 3 and 6 months of intervention.
  Body fat mass change assessed by difference in fat mass (%) comparing 3 and 6 months visits with respect to baseline.
Fat-free mass change. | After 3 and 6 months of intervention.
  Fat-free mass change assessed by difference in fat free-mass (%) comparing 3 and 6 months visits with respect to baseline.
Visceral fat mass change. | After 3 and 6 months of intervention.
  Visceral fat mass change assessed by difference in visceral fat mass (kg and %) comparing 3 and 6 months visits with respect to baseline.

SECONDARY OUTCOMES:
Total cholesterol change. | After 3 and 6 months of intervention.
  Total cholesterol change assessed by difference in fasting total cholesterol concentration (mg/dL and %) comparing 3 and 6 months visits with respect to baseline.
LDL cholesterol change. | After 3 and 6 months of intervention.
  Total LDL cholesterol change assessed by difference in fasting LDL cholesterol concentration (mg/dL and %) comparing 3 and 6 months visits with respect to baseline.
HDL cholesterol change. | After 3 and 6 months of intervention.
  HDL cholesterol change assessed by difference in fasting HDL cholesterol concentration (mg/dL and %) comparing 3 and 6 months visits with respect to baseline.
Triglycerides change. | After 3 and 6 months of intervention.
  Triglycerides change assessed by difference in fasting triglycerides concentration (mg/dL and %) comparing 3 and 6 months visits with respect to baseline.

OTHER OUTCOMES:
C-reactive protein change. | After 3 and 6 months of intervention.
  C-reactive protein change assessed by difference in fasting C-reactive protein concentration (mg/dL and %) comparing 3 and 6 months visits with respect to baseline.
Liver enzymes change. | After 3 and 6 months of intervention.
  Liver enzymes (GGT, GOT and GPT) change assessed by difference in fasting liver enzymes concentration (U/L and %) comparing 3 and 6 months visits with respect to baseline.
Uric acid change. | After 3 and 6 months of intervention.
  Uric acid change assessed by difference in fasting uric acid concentration (mg/dL and %) comparing 3 and 6 months visits with respect to baseline.
GLP-1 change. | After 3 and 6 months of intervention.
  GLP-1 change assessed by difference in fasting GLP-1 concentration (pg/mL and %) comparing 3 and 6 months visits with respect to baseline.
GIP change. | After 3 and 6 months of intervention.
  GIP change assessed by difference in fasting GIP concentration (pg/mL and %) comparing 3 and 6 months visits with respect to baseline.
IL-6 change. | After 3 and 6 months of intervention.
  IL-6 change assessed by difference in fasting IL-6 concentration (pg/mL and %) comparing 3 and 6 months visits with respect to baseline.
Leptin change. | After 3 and 6 months of intervention.
  Leptin change assessed by difference in fasting leptin concentration (pg/mL and %) comparing 3 and 6 months visits with respect to baseline.
MCP1 change. | After 3 and 6 months of intervention.
  MCP1 change assessed by difference in fasting MCP1 concentration (pg/mL and %) comparing 3 and 6 months visits with respect to baseline.
TNF-alpha change. | After 3 and 6 months of intervention.
  TNF-alpha change assessed by difference in fasting TNF-alpha concentration (pg/mL and %) comparing 3 and 6 months visits with respect to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Investigación Sanitaria Aragón, Hospital Universitario Miguel Servet, Universidad de Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodrigo-Carbo C, Madinaveitia-Nisarre L, Perez-Calahorra S, Gracia-Rubio I, Cebollada A, Galindo-Lalana C, Mateo-Gallego R, Lamiquiz-Moneo I. Low-calorie, high-protein diets, regardless of protein source, improve glucose metabolism and cardiometabolic profiles in subjects with prediabetes or type 2 diabetes and overweight or obesity. Diabetes Obes Metab. 2025 Jan;27(1):268-279. doi: 10.1111/dom.16013. Epub 2024 Oct 17. PMID 39420528